CLINICAL TRIAL: NCT05749172
Title: Effects of 8-weeks Strength Training on Strength Program, Power and Agility in Traceurs. A Randomized Controlled Trial
Brief Title: Effects of 8-weeks Strength Training on Strength Program, Power and Agility in Traceurs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: umairahamed0449
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group was provided with Strength training along with parkour routine training.
  Interventions: Other: Strength group
- Group B (Active Comparator): The control group was provided with parkour routine training
  Interventions: Other: Controlled group

INTERVENTIONS:
Other: Strength group — 4 sets of strength training exercises with 10 repetitions determined from ACSM two days a week, with a minimum of 72 hours between these days. In this exercise protocol, the movements of back squat, seated leg extension, seated leg curls, machine hip adductions, machine hip abductions, standing calf raises, back lat pulldowns, seated rows, bench press, incline bench press, biceps curls, triceps pushdowns, back press, back extension, pushup, pullup, squats and sit-ups will be performed.
  Arms: Group A
Other: Controlled group — Two hours of parkour training for two days a week.
  Arms: Group B

SUMMARY:
The goal of this Randomized controlled trial was to examine effects of 8-weeks strength training program on strength, power and agility in traceurs. The main question it aims to answer is:

• To determine the effects of 8-weeks strength training program in traceurs. Participants were a given consent form and after subjects read and sign the informed consent, they were included in study according to eligibility criteria. 2 groups were included in study, Strength Group with parkour routine training was applied on group A and the control group, group B was provided with parkour routine training. Outcome was measured through different outcome measure tools.

DETAILED DESCRIPTION:
The parkour is a physical activity that contains exceptional technique applications and requires a major number of jumps. The purpose of this study was to examine the effects of 8-week strength training on strength program, power, and agility in traceurs (parkour practitioners). Officially incorporated as a sport in the UK in 2017 but born in France almost 30 years ago. Parkour consists of practitioners finding a route through predominantly urban terrain, mastering various physical and psychological skills to overcome obstacles in the most efficient, effective way possible.

A randomized controlled trial will be performed in which total 16 traceurs will be observed for 8 weeks. The data was collected from Pakistan Parkour & Free running Academy in Quetta, Balochistan. Participants would be randomly divided into two balanced groups. One group was provided with parkour training sessions, and the other group was provided with both strength and parkour training sessions. The participants, who have done strength training along with the parkour trainings, apply 4 sets of strength training exercises with 10 repetitions determined from ACSM two days a week, with a minimum of 72 hours between these days. The control group was applied only two hours of parkour training for two days a week.

Aim of study was to observe effects of strength training in vertical jump heights at the end of the 8-week strength trainings comparison to the control group and that of the strength training. This study aids in learning of the vertical jump heights by including strength training programs with routine trainings, which is a central parameter for successful performance in traceurs, can enable the coaches and athletes to prepare a better training.

ELIGIBILITY:
Inclusion Criteria:

* Age (16-30years)
* Male traceurs
* Parkour participants had been involved in parkour practice for at least two years (2 times per week for a minimum of 2 hours per day) and did not have any bone, articular or muscular injuries in the previous 6 months.

Exclusion Criteria:

* Participants been involved in strength training before.
* Participants not been involved in parkour practice for minimum 2years.
* Participant who have injuries within previous 6 months.
* Participants who smokes or were taking medication.

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2023-02-18 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Vertical jump (power) | 8 weeks
  Vertical jump tests provide an effective measurement of power as an indirect measure of performance. Strength and conditioning professionals have long used performance tests such as the vertical jump to assess athletic ability, which helps them to identify athletes, strengths and weaknesses, chart and document progress, or assign positions and ranking to individuals. vertical jump testing is being used to measure the effectiveness of various training programs in developing explosive power, including strength training programs.
Agility t-test | 8 weeks
  The agility T-test may be a useful tool to assess athlete function and changes in performance during training and rehabilitation programs. The T-test is described as a measure of 4-directional agility and body control that evaluates the ability to change directions rapidly while maintaining balance without loss of speed.
Dynamic strength | 8 weeks
  The push-up test is a basic fitness test used by coaches, trainers, and athletes to assess upper body fitness and to monitor progress during strength and fitness training.
  The pull-up is a closed kinetic chain, multi-joint upper-body exercise that can improve an athlete's shoulder girdle strength, stability, and ability to produce high forces during pulling activities.
  The overhead squat test is a subjective screening assessment used to obtain a general indication of dynamic posture. The test identifies compensatory movements and considers muscles which could potentially be overactive or underactive with the intention of addressing these muscle imbalances.

CONTACTS AND LOCATIONS:
Overall Officials: Umair Ahmed, Principal Investigator — Ripahah International University
Locations (1):
- Pakistan Parkour & Freerunning Academy in Quetta, Balochistan, Quetta, Balochistan, Pakistan